CLINICAL TRIAL: NCT00001324
Title: CNS Control of Human Movement: H215O PET Studies
Brief Title: PET Scan to Study Brain Control of Human Movement
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920119; 92-N-0119
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2000-03

CONDITIONS: Ataxia; Cerebrovascular Accident; Healthy; Movement Disorder; Tremor
Keywords: Ataxia; Brain; Motor Learning; Parkinson's Disease; Physiology; Positron Emission Tomography; Stroke; Tremor; Voluntary and Involuntary Movement Physiology; Movement Disorders; Normal Volunteer
MeSH Terms: conditions — Ataxia; Stroke; Movement Disorders; Tremor; Parkinson Disease

SUMMARY:
Positron Emission Tomography (PET) is a technique used to investigate activity in areas of the brain. The PET technique allows researchers to study the normal processes in the brain (central nervous system) of normal individuals and patients with neurologic illnesses without physical / structural damage to the brain.

When a region of the brain is active, it uses more fuel in the form of oxygen and sugar (glucose). As the brain uses more fuel it produces more waste products, carbon dioxide and water. Blood carries fuel to the brain and waste products away from the brain. As brain activity increases, blood flow to and from the area of activity also increases. This is known as regional cerebral blood flow (rCBF). Knowing these facts, researchers can use radioactive water (H215O) and PET scans to observe what areas of the brain are receiving more blood flow.

In this study researchers plan to investigate the changes in regional cerebral blood flow (rCBF) as patients participate in different activities. The activities are designed to stimulate the areas of the brain responsible for voluntary motor activity and sensation. By comparing the results of PET scans performed in different conditions, researchers can locate regions of the brain responsible for specific tasks.

This study should provide new information about voluntary movements in humans and the preparation involved in controlling them.

DETAILED DESCRIPTION:
The main purpose of the studies presented in this protocol is to investigate the physiology of motor control in health as well as the pathophysiological modifications taking place during disease. To this end, we will investigate changes in regional cerebral blood flow (rCBF) as an index of regional neuronal activity, associated with various motor and sensory tasks using Positron Emission Tomography (PET). The rCBF will be obtained by measuring the distribution of the cerebral radioactivity during emission scans following the intravenous bolus injection of 15O-labeled water. The very short half-life of 15O (2 minutes) allows us to measure rCBF repeatedly under different task conditions (see methodology and experimental procedures). With the comparison between PET scans performed in different conditions, we can detect the specific task-related activated regions. PET images will be coregistered to high resolution Magnetic Resonance Images (MRI) to get more accurate anatomical information regarding the activated areas. The results will be correlated with that from other physiological approaches including Electroencephalography (EEG), Transcranial Magnetic Stimulation (TMS), functional Magnetic Resonance Imaging (fMRI), and Magnetic Resonance Spectroscopy (MRS). These studies should provide new information not only about the executive component of the voluntary movements in humans but also the different organizational aspects of the preparatory processes that control them.

ELIGIBILITY:
Patients with movement disorder and normal volunteers.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 510
Dates: Start 1992-03; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Deiber MP, Ibanez V, Honda M, Sadato N, Raman R, Hallett M. Cerebral processes related to visuomotor imagery and generation of simple finger movements studied with positron emission tomography. Neuroimage. 1998 Feb;7(2):73-85. doi: 10.1006/nimg.1997.0314. PMID 9571132
- [Background] Catalan MJ, Honda M, Weeks RA, Cohen LG, Hallett M. The functional neuroanatomy of simple and complex sequential finger movements: a PET study. Brain. 1998 Feb;121 ( Pt 2):253-64. doi: 10.1093/brain/121.2.253. PMID 9549504
- [Background] Deiber MP, Wise SP, Honda M, Catalan MJ, Grafman J, Hallett M. Frontal and parietal networks for conditional motor learning: a positron emission tomography study. J Neurophysiol. 1997 Aug;78(2):977-91. doi: 10.1152/jn.1997.78.2.977. PMID 9307128